CLINICAL TRIAL: NCT02128282
Title: A Phase I/II Study of CX-4945 in Combination With Gemcitabine and Cisplatin in the Frontline Treatment of Patients With Cholangiocarcinoma
Brief Title: Study of CX-4945 in Combination With Gemcitabine and Cisplatin for Frontline Treatment of Cholangiocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Senhwa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S4-13-001
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Bile duct cancer; Biliary tract cancer
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms; Biliary Tract Neoplasms | interventions — silmitasertib; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Escalation CX-4945 plus Cis/Gem (Experimental): CX-4945 capsules at the combination MTD on Days 0, 1 and 2, and Days 7, 8 and 9.
  PLUS Cisplatin 25 mg/m.sq. by IV infusion on Days 1 and 8. PLUS Gemcitabine 1,000 mg/m.sq. by IV infusion on Days 1 and 8. On a 21-day cycle.
  Interventions: Drug: CX-4945; Drug: Cisplatin; Drug: Gemcitabine
- Cisplatin plus Gemcitabine (Active Comparator): Cisplatin 25 mg/m.sq. by IV infusion on Days 1 and 8. PLUS Gemcitabine 1,000 mg/m.sq. by IV infusion on Days 1 and 8. On a 21-day cycle.
  Interventions: Drug: Cisplatin; Drug: Gemcitabine
- 10-day CX-4945 plus Cis/Gem (Experimental): CX-4945 capsules at 1000mg/BID, 10-day continuous dosing (Day 0 through Day 9). PLUS Cisplatin 25 mg/m.sq. by IV infusion on Days 1 and 8. PLUS Gemcitabine 1,000 mg/m.sq. by IV infusion on Days 1 and 8. On a 21-day cycle.
  Interventions: Drug: CX-4945; Drug: Cisplatin; Drug: Gemcitabine
- 21-day CX-4945 plus Cis/Gem (Experimental): CX-4945 capsules at 1000mg/BID, 21-day continuous dosing PLUS Cisplatin 25 mg/m.sq. by IV infusion on Days 1 and 8. PLUS Gemcitabine 1,000 mg/m.sq. by IV infusion on Days 1 and 8. On a 21-day cycle.
  Interventions: Drug: CX-4945; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: CX-4945 — API powder-in-capsule in 200 mg strength.
  Arms: 10-day CX-4945 plus Cis/Gem; 21-day CX-4945 plus Cis/Gem; Escalation CX-4945 plus Cis/Gem
Drug: Cisplatin — 25 mg/m.sq. administered by IV infusion on Days 1 and 8 of a 21-day cycle.
  Other Names: Platinol
Drug: Gemcitabine — 1,000 mg/m.sq. administered by IV infusion on Days 1 and 8 of a 21-day cycle.
  Other Names: Gemzar

SUMMARY:
This study considers the safety and tolerability of increasing doses of CX-4945 in combination with gemcitabine plus cisplatin to determine the maximum tolerated dose (MTD) and the recommended Phase II dose (RP2D), followed by a randomized study that compares antitumor activity in cholangiocarcinoma patients receiving the standard of care gemcitabine plus cisplatin versus CX-4945 at the combination RP2D with gemcitabine plus cisplatin.

DETAILED DESCRIPTION:
Protein kinase CK2 is a constitutively active serine/threonine kinase with a long history as a pro-survival, anti-apoptotic kinase. Given the wide spread overexpression of CK2 in multiple cancers and its role in multiple non-oncogenic processes required to sustain the cancer phenotype, a selective inhibitor of CK2 is an attractive targeted approach to treating cancer.

CX-4945 is a tetracyclic, small molecule carboxylate acid salt that exhibits potent and highly selective inhibition of CK2. Protein kinase CK2 is also known to play an important role in the DNA damage repair mechanisms of cancer cells, and this study of CX-4945 in combination with gemcitabine plus cisplatin will determine if inhibition of CK2, in conjunction with the use of chemotherapy drugs, will result in improved clinical outcomes for patients with non-resectable cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an unresectable hepatobiliary mass or metastatic disease (consistent with cholangiocarcinoma, as evidenced by histology or cytology (augmented by fluorescence in situ hybridization (FISH) where appropriate), for which treatment with gemcitabine plus cisplatin is intended. Intrahepatic and extrahepatic cholangiocarcinoma patients may be enrolled.
* For patients enrolled in the Dose Escalation Phase, one or more tumors measurable on radiograph or CT scan, or evaluable disease defined as non-measurable lesions per RECIST v. 1.1 (e.g., malignant ascites). All patients enrolled to the Randomized Study Phase must have measurable disease only.
* Laboratory data as specified below:

  * Hematology: Absolute neutrophil count (ANC) >1,500 cells/mm3, platelet count >100,000 cells/ mm.cu. and hemoglobin > 9 g/dL
  * Hepatic: bilirubin <1.5 X Upper Limit of Normal (ULN); alkaline phosphatase (ALP), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5.0 X ULN
  * Renal: serum creatinine within normal limits (WNL), defined as within 25% of the institution's stated reference range, or a calculated creatinine clearance >45 mL/min/1.73 m. sq. for patients with abnormal, increased, creatinine levels.
  * Coagulation: International Normalized Ratio (INR) < 1.5 times normal, activated Partial Thromboplastin Time (aPTT) < 1.5 times normal. Patients receiving therapeutic doses of anticoagulant therapy may be considered eligible for the trial if INR and aPTT are within the acceptable therapeutic limits for the institution.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 1.

Exclusion Criteria:

* A history of prior systemic treatment with gemcitabine or cisplatin. At least six months must have elapsed if gemcitabine or cisplatin was administered in an adjuvant treatment setting. Patients enrolled in the Expansion Cohort, Exploratory Cohorts, and the Randomized Phase must not have received prior systemic chemotherapies, including chemoradiation therapy for cholangiocarcinoma.
* Seizure disorders requiring anticonvulsant therapy.
* Known brain metastases (unless previously treated and well controlled for a period of at least 3 months).
* Major surgery other than diagnostic surgery, within 4 weeks prior to the first dose of test drug, minor surgery including diagnostic surgery within 2 weeks (14 days) excluding central IV port placements and needle aspirate/core biopsies. Radio frequency ablation or transcatheter arterial chemoembolization within 6 weeks prior to the first dose of test drug.
* Treatment with radiation therapy or surgery within one month prior to study entry.
* Treatment with chemotherapy or investigational drugs within 21 days prior to the screening visit. Acute toxicities from prior therapy must have resolved to Grade ≤ 1 above baseline.
* Patients with a history of another malignancy within 3 years of the baseline visit. (Patients with cutaneous carcinomas or in-situ carcinomas will be considered for study entry on a case-by-case basis).
* Concurrent severe or uncontrolled medical disease (i.e., systemic infection, diabetes, hypertension, coronary artery disease, congestive heart failure).
* Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral (A, B or C) hepatitis which would not permit the patient to be managed according to the protocol.
* Difficulty with swallowing or an active malabsorption syndrome.
* Chronic diarrhea (excess of 2-3 stools/day above normal frequency).
* Gastrointestinal diseases including ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of gastric or small bowel surgery involving any extent of gastric or small bowel resection.
* Clinically significant bleeding event within the last 3 months, unrelated to trauma, or underlying condition that would be expected to result in a bleeding diathesis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of CX-4945 when used in combination with gemcitabine plus cisplatin. (Phase 1) | Cycle 1, 1 Full cycle up to twenty-one (21) days
  The Maximum Tolerated Dose of CX-4945 will be determined from safety observations during the first cycle, as the CX-4945 dose is escalated in cohorts of three patients in combination with standard gemcitabine plus cisplatin.
Comparison of the Progression-free survival (PFS) between the test and the control arms using Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 (Phase 2) | From date of randomization to date of progression or death from any cause up to 52 weeks.
  Tumor measurements will be compared to baseline every six weeks, and the PFS will be determined using RECIST v. 1.1.
Recommended Phase II dose (RP2D) and schedule of CX-4945 in combination with gemcitabine plus cisplatin (Phase I) | Cycle 1, 1 Full cycle up to twenty-one (21) days
  The recommended Phase II dose and schedule of CX-4945 will be determined from safety observations during the first cycle, as the CX-4945 dose is administered 1000mg BID in 10-day continuous or 21-day continuous cohorts in combination with standard gemcitabine plus cisplatin.

SECONDARY OUTCOMES:
Comparison of the Overall Response Rate (ORR) between the test and the control arms using Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 | From date of randomization to date of progression or death from any cause up to 52 weeks.
  Tumor measurements will be compared to baseline, and the ORR will be determined using RECIST v. 1.1
Comparison of the number of patient who transition to surgical resection | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The number of patients in the chemotherapy arm versus CX-4945 plus chemotherapy arm who transition to surgical resection will be compared.
Comparison of the Overall Survival (OS) between the test and the control arms | From date of randomization to date of death from any cause up to 52 weeks.
  Time to event is observed during treatment and followed up every 3 months after patient withdraw from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Borad, M.D., Principal Investigator — Mayo Clinic
Locations (16):
- United States (6):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Colorado- Denver, Aurora, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Tyler, Tyler, Texas
- South Korea (4):
  - Asan Medical Center, Seoul, Songpa-gu
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Taiwan (6):
  - Chang-Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospitals, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital - Linkou Branch, Taoyuan

IPD SHARING:
Plan to Share IPD: No